CLINICAL TRIAL: NCT01889732
Title: The Effectiveness Evaluation of Rotational Thromboelastometry(ROTEM) for Predicting Postoperative Bleeding in Cardiac Surgical Patients Using a Gray Zone Approach : A Preliminary Retrospective Study
Brief Title: A Gray Zone Approach of Rotational Thromboelastometry for Predicting Postoperative Bleeding in Cardiac Surgical Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: SMC 2013-05-060
Record Dates: First submitted 2013-06-20; First posted 2013-06-28 (Estimated); Last update posted 2013-06-28 (Estimated); Status verified 2013-06

CONDITIONS: Other Functional Disturbances Following Cardiac Surgery; Postoperative Hemorrhage; Coagulation Defect; Bleeding
MeSH Terms: conditions — Postoperative Hemorrhage; Hemostatic Disorders; Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- ROTEM
  Interventions: Device: ROTEM

INTERVENTIONS:
Device: ROTEM

SUMMARY:
Rotational thromboelastometry (ROTEM) is reliable point of care management of coagulation disorder undergoing surgery. Recently, there are some reports about prediction of perioperative bleeding using ROTEM. But, the effectiveness of ROTEM for predict bleeding and improve outcomes is still debate. In this retrospective study, the investigators will compare immediate postoperative bleeding with ROTEM parameters using a Gray zone approach, and access the reliability of ROTEM for prediction of bleeding after cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* cardiac surgical patients using Cardiopulmonary bypass

Exclusion Criteria:

* known coagulation disorder
* Using deep hypothermic circulatory arrest
* Using partial cardiopulmonary bypass

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: elective cardiac surgical patient age 20-80years
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2013-06; Primary Completion 2013-08 (Estimated); Study Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
early postoperative bleeding(chest tube drainage) | postoperative bleeding during 6hrs.
  primary outcome is Chest tube drainage(blood volume) during 6hrs.

CONTACTS AND LOCATIONS:
Overall Officials: jonghwan lee, MD, PhD, Principal Investigator — Samsung Medical Center; eunhee kim, MD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea